CLINICAL TRIAL: NCT02236442
Title: Therapeutic Management of Acute Cephalalgia Before and After Use of a Therapeutic Protocol in Emergency Department
Brief Title: Protocol to Ease Acute Cephalalgia in Emergency-department
Acronym: PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00973-44
Record Dates: First submitted 2014-08-07; First posted 2014-09-10 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Cephalalgia
Keywords: Cephalalgia; Headache; Migraine; Pain; Global; Treatment; Oxygen; Emergency; Treatment of cephalalgia in emergency department
MeSH Terms: conditions — Headache; Migraine Disorders; Pain; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): First arm : Passive recording head pain, linked symptoms, treatment used and diagnosis.
- After protocol recommendation care (Experimental): Recording head pain, linked symptoms, treatment used and diagnosis after intervention that is recommendation to use global headache treatment protocol
  Interventions: Other: Recommendation to use global headache treatment protocol

INTERVENTIONS:
Other: Recommendation to use global headache treatment protocol — The global treatment protocol is :
  1. Put the patient in a quiet spot, ideally an individual room. Avoid waiting in the corridor
  2. Lay down the patient on the stretcher. Avoid waiting on a seat or a chair.
  3. Provide a sound-proof helmet to the patient.
  4. Provide a light-blocking google to the patient.
  5. If judged necessary by the physician in charge of the patient, administer oxygen therapy, 15 liter per minute, during 15 minutes.
  6. If judged necessary by the physician in charge of the patient, administer analgesic treatment adapted to the etiology of the cephalalgia as described :
  Migraine : acetylsalicilyc acid + metoclopramide or nonsteroidal anti inflammatory or paracetamol or triptan.
  Tension headache : nonsteroidal anti inflammatory or paracetamol. Avoid methylmorphine or tramadol if possible.
  Cluster headache : Intravenous or nasal spray sumatriptan and oxygen therapy.
  Other etiology : Treatment left at the discretion of the physician in charge of the patient.
  Arms: After protocol recommendation care

SUMMARY:
The purpose of this study is to determine if the use of a therapeutic and global protocol to relieve cephalalgia is helpful in the emergency department of Grenoble University Hospital.

DETAILED DESCRIPTION:
Cephalalgia is a very common symptom that justifies daily appointment in emergency department.

Analgesic support, and especially use of oxygen and care of associated symptoms as nausea, photophobia or phonophobia, is very dependent on the physician.

The aim of this study is to evaluate the impact of a global analgesic protocol of cephalalgia in emergency department.

The investigators included 200 patients aged of 18 up to 55 years old coming in emergency department for headache. Pain (Visual analogic scale), nausea, photo or phonophobia are recorded each 15 minutes by the patient by using a self-assessment questionnaire. The final diagnosis is recorded by the physician in charge of patient, using International Headache Society criteria.

First 100 patients(group 1) receive usual care.

For the last 100 patients (group 2), physician in charge of patients are incited to use a formal protocol that include: putting the patient in a quiet spot, laying down on a stretcher, providing sound proof helmet and light blocking google, administering oxygen therapy 15 l/min during 15 min, and administering etiological headache adapted medication following learned society guidelines.

Comparison of the data of this 2 groups shall help us to see if the investigators actual analgesic support of cephalalgia is efficient, and if it can be improved by this global analgesic protocol.

ELIGIBILITY:
Inclusion Criteria:

* Complain about cephalalgia
* Age 28 to 55 years.

Exclusion Criteria:

* Fever > 38,0 °C
* History of breath disease, long term use of oxygen therapy, chronic obstructive pulmonary disease, dyspnea
* History of cranial traumatism, heart attack, cerebrovascular accident <3 month
* Inability to read or understand french.
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 1 hour after treatment
  "Clinical improvement" is defined as "Reduction of at least 50% of quantified pain 1 hour after treatment Comparison of proportion of "clinical improvement" between the 2 groups.

SECONDARY OUTCOMES:
Pain score on the visual analog scale | 1 hour after treatment
  Measure of amount of pain by recording quantified pain evaluation each 15 minutes. Analysis by ANOVA (Analysis of Variance).
  Comparison between the 2 groups.
Pain depending on the kind of cephalalgia | 1 hour after treatment
  Research of interaction between the occurrence of the "clinical improvement" and the cephalalgia diagnosis (Migraine, tensive headache, cluster headache, secondary headache...).
Impact of different kind of analgesic therapeutic | 1 hour after treatment
  Research of interaction between the occurrence of "clinical improvement" and the use of specific therapeutic strategy ( Restful position, calm environment, wearing opaque glasses, soundproof headset, oxygen therapy, other medication, ...)
Length of the hospitalization in emergency department | Duration of hospitalisation in emergency department stay, an expected average of 6 hours
  Evaluation of the length of the hospitalization in emergency department. Comparison between the 2 groups
Time required before medication | Time of administration of first medication, an expected average of 30 minutes
  Evaluation of the length of time before first administration of analgesic treatment.
  Comparison between the 2 groups
Hospitalisation requirement | Exit of emergency department, an expected average of 6 hours
  Evaluation of hospitalisation requirement at the exit of emergency department.
  Comparison between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mirebeau, Resident, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, Isere, France

REFERENCES:
- [Background] Rasmussen BK, Jensen R, Schroll M, Olesen J. Epidemiology of headache in a general population--a prevalence study. J Clin Epidemiol. 1991;44(11):1147-57. doi: 10.1016/0895-4356(91)90147-2. PMID 1941010
- [Background] Friedman BW, Grosberg BM. Diagnosis and management of the primary headache disorders in the emergency department setting. Emerg Med Clin North Am. 2009 Feb;27(1):71-87, viii. doi: 10.1016/j.emc.2008.09.005. PMID 19218020
- [Background] Haque B, Rahman KM, Hoque A, Hasan AT, Chowdhury RN, Khan SU, Alam MB, Habib M, Mohammad QD. Precipitating and relieving factors of migraine versus tension type headache. BMC Neurol. 2012 Aug 25;12:82. doi: 10.1186/1471-2377-12-82. PMID 22920541
- [Background] Cohen AS, Burns B, Goadsby PJ. High-flow oxygen for treatment of cluster headache: a randomized trial. JAMA. 2009 Dec 9;302(22):2451-7. doi: 10.1001/jama.2009.1855. PMID 19996400
- [Background] Ozkurt B, Cinar O, Cevik E, Acar AY, Arslan D, Eyi EY, Jay L, Yamanel L, Madsen T. Efficacy of high-flow oxygen therapy in all types of headache: a prospective, randomized, placebo-controlled trial. Am J Emerg Med. 2012 Nov;30(9):1760-4. doi: 10.1016/j.ajem.2012.02.010. Epub 2012 May 3. PMID 22560101
- [Background] Matharu M. Cluster headache. BMJ Clin Evid. 2010 Feb 9;2010:1212. PMID 21718584
- [Background] B. D VEYSMAN, et al. Oxygen Therapy for the tratment of undifferentiated headache in the emergency department. ClinicalTrials.gov, NCT00856232